CLINICAL TRIAL: NCT03376126
Title: Minimally-Invasive Isolated Limb Perfusion
Acronym: MI-ILP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate professor, Sahlgrenska University Hospital
Other Study IDs: MI-ILP
Record Dates: First submitted 2017-12-08; First posted 2017-12-18 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Isolated Limb Perfusion
Keywords: isolated limb perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MI-ILP
  Interventions: Other: Minimal-invasive isolated limb perfusion

INTERVENTIONS:
Other: Minimal-invasive isolated limb perfusion — Minimal-invasive isolated limb perfusion

SUMMARY:
The aim is to analyse feasibility of a minimally-invasive isolated limb perfusion.

DETAILED DESCRIPTION:
Isolated limb perfusion (ILP) and isolated limb infusion (ILI) are treatment options for patients with in-transit metastases of melanoma and locally advanced extremity sarcomas. There are several advantages for each method, but if the well-established effects of ILP could be combined to the minimally invasive approach of ILI, the results could be maximized and adverse events, related to open approach, minimized.

A new method for vascular approach (MI-ILP) will be evaluated in a phase I feasibility study. Percutaneous vascular access of the ipsilateral side will be performed by ultrasound guided technique and connected to an extracorporeal oxygenation system. Perfusion will be conducted in the same way as for open ILP. Outcomes, technical details and complications will be recorded prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. The patient scheduled for treatment with isolated hyperthermic perfusion
2. Age over 18 years.
3. Signed informed consent

Exclusion Criteria:

1. Re-perfusion
2. Lymph node metastases
3. Severe atherosclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for isolated limb perfusion.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Conversion to open surgery | 1 day
  Number of minimal-invasive procedure that will be converted to open surgery (per cent)

SECONDARY OUTCOMES:
Response | 3 months
  Clinical response rate according to WHO criteria.
Complications | 30 days
  Complications according to Clavien-Dindo

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No